CLINICAL TRIAL: NCT00002095
Title: A Randomized, Double-Blind Study of the Efficacy and Safety of Oral Ganciclovir for the Prevention of CMV Disease in People Infected With the Human Immunodeficiency Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 059D; ICM 1654
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-11

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: Ganciclovir; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To evaluate the efficacy of oral ganciclovir in preventing progression to cytomegalovirus (CMV) disease (e.g., CMV retinitis, gastrointestinal CMV disease) in CMV-infected people with HIV infection and CD4 lymphocyte counts <= 100 cells/mm3. To evaluate the efficacy of this drug in reducing morbidity associated with coinfection by both CMV and HIV.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Topical or ophthalmic nucleoside analogs.

Patients must have:

* Confirmation of HIV infection.
* Documented CMV infection.
* No past or present CMV disease (e.g., retinitis, colitis, esophagitis).
* Adequate visualization of the retina of both eyes by ophthalmologist.
* CD4 count <= 50 cells/mm3 (in patients WITHOUT a history of an AIDS-defining opportunistic infection or chronic gynecologic infection) OR CD4 count <= 100 cells/mm3 (in patients WITH a history of an AIDS-defining opportunistic infection or chronic gynecologic infection).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Presence of gastrointestinal disease or symptoms not controlled with medications (e.g., persistent nausea, abdominal pain or persistent diarrhea within the past 4 weeks that is not controllable with medication).
* Inability to comply with protocol.

Concurrent Medication:

Excluded:

* The following nucleoside analogs:
* IV ganciclovir, IV acyclovir for more than 2 weeks total duration, oral acyclovir at doses > 1000 mg/day, vidarabine, amantadine hydrochloride, cytarabine, idoxuridine.
* FIAU, FIAC, foscarnet, CMV hyperimmune globulin, IV immune globulin, CMV monoclonal antibody, HPMPC.
* Imipenem-cilastatin (Primaxin).

Patients with the following prior condition are excluded:

History of hypersensitivity to acyclovir.

Prior Medication:

Excluded within the past 60 days:

Ganciclovir, foscarnet, FIAC, FIAU, CMV hyperimmune globulin, CMV monoclonal antibody, or HPMPC.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - East Bay AIDS Ctr, Berkeley, California
  - Kraus - Beer Med Group, Los Angeles, California
  - UCSD, San Diego, California
  - Davies Med Ctr / c/o HIV Institute, San Francisco, California
  - Mount Zion Med Ctr, San Francisco, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Community Research Initiative, Coral Gables, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr / Rush Med Coll, Chicago, Illinois
  - Beth Israel Hosp, Boston, Massachusetts
  - Kaplan Cancer Ctr / New York Univ Med Ctr, New York, New York
  - St Lukes - Roosevelt Hosp Ctr, New York, New York
  - Cornell Univ Med College / New York Hosp, New York, New York
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Univ of Pittsburgh / Graduate School of Public Health, Pittsburgh, Pennsylvania
  - Oak Lawn Physicians Group, Dallas, Texas
  - Infectious Diseases Association of Houston, Houston, Texas

REFERENCES:
- [Background] Spector SA, McKinley GF, Lalezari JP, Samo T, Andruczk R, Follansbee S, Sparti PD, Havlir DV, Simpson G, Buhles W, Wong R, Stempien M. Oral ganciclovir for the prevention of cytomegalovirus disease in persons with AIDS. Roche Cooperative Oral Ganciclovir Study Group. N Engl J Med. 1996 Jun 6;334(23):1491-7. doi: 10.1056/NEJM199606063342302. PMID 8618603